CLINICAL TRIAL: NCT00000848
Title: The Antiviral Effect of Switching From Hard Capsule Saquinavir (SQVhc) to the Soft Gelatin Capsule of Saquinavir (SQVsc) Versus Switching to Indinavir (IDV) After 1 Year of Saquinavir Use
Brief Title: The Anti-HIV Effects of Saquinavir Soft Gelatin Capsules Versus Indinavir in Patients Who Have Used Saquinavir Hard Gelatin Capsules for One Year
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 333; 11305 (Registry Identifier: DAIDS ES)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Administration, Oral; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Antiviral Agents; HIV Protease Inhibitors; Biological Markers; Indinavir; Viremia; RNA, Viral; Saquinavir
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Viremia | interventions — Indinavir; Saquinavir

INTERVENTIONS:
Drug: Indinavir sulfate
Drug: Saquinavir

SUMMARY:
To determine, in HIV-infected patients, whether switching to a new soft gelatin capsule formulation of saquinavir or to indinavir following prolonged use of the original hard capsule formulation of saquinavir results in an acute decrease in plasma HIV RNA.

Resistance to anti-HIV agents occurs with increasing duration of use. In vitro studies have shown that cross-resistance occurs among protease inhibitors, although no clinical trials have been conducted to examine antiretroviral activity with sequential use of protease inhibitors or to determine whether saquinavir resistance can be overcome with higher concentrations of the drug.

DETAILED DESCRIPTION:
Resistance to anti-HIV agents occurs with increasing duration of use. In vitro studies have shown that cross-resistance occurs among protease inhibitors, although no clinical trials have been conducted to examine antiretroviral activity with sequential use of protease inhibitors or to determine whether saquinavir resistance can be overcome with higher concentrations of the drug.

Patients who are currently receiving hard capsule saquinavir are randomized to continue receiving hard capsule saquinavir or to switch to soft gelatin capsule saquinavir or indinavir. At week 8, patients receiving the hard capsule formulation will switch to open-label indinavir for weeks 8-24. Patients on the other two arms will remain on their assigned regimen for the entire 24 weeks unless they have no virologic response by week 8, in which case they will be crossed-over to open-label therapy with the alternative drug (i.e., either soft gelatin capsule saquinavir or indinavir).

AS PER AMENDMENT 12/23/96: Viral RNA from weeks 16 and 24 will be assayed in batch after week 24. Patients who exhibit an antiviral response based on this assay will be allowed to continue their current drug assignment for a total of 12 months.

AS PER AMENDMENT 5/7/97: Based on an interim analysis performed after 72 patients had completed 8 weeks of therapy, the study was closed as of March 7, 1997. Patients currently enrolled may stop their participation in the trial and seek other anti-retroviral therapies or may continue on study. Patients on hard capsule saquinavir who remain on study will be switched to indinavir at 8 weeks. Patients on soft gel capsule saquinavir may switch immediately to indinavir or, when results of HIV RNA and CD4 cell counts are available, may choose to switch to indinavir or remain on soft gel capsule saquinavir. Patients receiving indinavir will continue that agent. Follow-up for all patients will end on 7/4/97.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Required:

* PCP prophylaxis if CD4 count <= 200 cells/mm3.

Allowed:

* Intralesional therapy for KS.
* Vitamins.
* Nucleoside RT inhibitors, provided regimen remains stable for first 8 weeks of study.

Concurrent Treatment:

Allowed:

* Acupuncture.
* Visualization techniques.

Patients must have:

* HIV infection.
* Prior hard capsule saquinavir at 1800 mg/day for more than 1 year.

Prior Medication:

Allowed:

* Prior saquinavir.
* Prior antiretrovirals, excluding protease inhibitors other than saquinavir.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Psychological condition or medical instability that would interfere with study evaluation or procedures.

AS PER AMENDMENT 5/7/97:

* Active tuberculosis.

Concurrent Medication:

Excluded:

* Protease inhibitors other than study drugs.
* Non-nucleoside RT inhibitors.
* Interferon.
* Interleukins.
* GM-CSF.
* HIV vaccines.
* Systemic cytotoxic chemotherapy.
* Investigational drugs other than study medications.
* Rifabutin.
* Rifampin.
* Midazolam.
* Triazolam.
* Ketoconazole.
* Delavirdine.
* Cisapride.
* Terfenadine.
* Astemizole.

AS PER AMENDMENT 5/7/97:

* Nevirapine.

Patients with the following prior conditions are excluded:

* Unexplained fever > 38.5 C for any 7 days within 30 days prior to study entry.
* Diarrhea persisting for 15 days within 30 days prior to study entry.

Prior Medication:

Excluded:

* Any prior protease inhibitor other than saquinavir.

Excluded within the past 2 months.

* Change in antiretroviral regimen.
* Systemic chemotherapy for KS.

Excluded within the past month:

* Non-nucleoside RT inhibitors.
* Interferons.
* Interleukins.
* HIV vaccines.
* Experimental therapies.

Excluded within the past 2 weeks:

* Rifabutin.
* Cisapride.
* Terfenadine.
* Astemizole.
* Midazolam.
* Triazolam.
* Oral ketoconazole.
* Delavirdine.
* Acute therapy for infection or other medical illness.

Active substance abuse that would interfere with study evaluation or procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Study Completion 1998-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Para MF, Study Chair; Collier A, Study Chair; Coombs R, Study Chair
Locations (16):
- United States (16):
  - Stanford CRS, Palo Alto, California
  - Ucsf Aids Crs, San Francisco, California
  - Harbor-UCLA Med. Ctr. CRS, Torrance, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Univ. of Miami AIDS CRS, Miami, Florida
  - Northwestern University CRS, Chicago, Illinois
  - Rush Univ. Med. Ctr. ACTG CRS, Chicago, Illinois
  - Massachusetts General Hospital ACTG CRS, Boston, Massachusetts
  - Washington U CRS, St Louis, Missouri
  - St. Louis ConnectCare, Infectious Diseases Clinic, St Louis, Missouri
  - SUNY - Buffalo, Erie County Medical Ctr., Buffalo, New York
  - Beth Israel Med. Ctr. (Mt. Sinai), New York, New York
  - NY Univ. HIV/AIDS CRS, New York, New York
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - The Ohio State Univ. AIDS CRS, Columbus, Ohio
  - University of Washington AIDS CRS, Seattle, Washington

REFERENCES:
- [Background] Saquinavir update. Treat Rev. 1997 Aug;(No 25):6. PMID 11364616
- [Background] Saquinavir switch study stopped. Treat Rev. 1997 Apr;(No 24):6. PMID 11364285
- [Background] Gilden D. Spring cleaning in trial land. GMHC Treat Issues. 1997 Mar;11(3):4-7. PMID 11364275
- [Background] Para MF, Coombs R, Collier A, Glidden D, Bassett R, Duff F, Boucher C, Leavitt RY, Condra J, Pettinelli C. Relationship of baseline genotype to RNA response in ACTG 333 after switching from long term saquinavir (SQVhc) to indinavir (IDV) or saquinavir soft gelatin capsule (SQVsgc). Conf Retroviruses Opportunistic Infect. 1998 Feb 1-5;5th:175 (abstract no 511)
- [Background] Sevin AD, DeGruttola V, Nijhuis M, Schapiro JM, Foulkes AS, Para MF, Boucher CA. Methods for investigation of the relationship between drug-susceptibility phenotype and human immunodeficiency virus type 1 genotype with applications to AIDS clinical trials group 333. J Infect Dis. 2000 Jul;182(1):59-67. doi: 10.1086/315673. Epub 2000 Jul 6. PMID 10882582
- [Background] Para MF, Glidden DV, Coombs RW, Collier AC, Condra JH, Craig C, Bassett R, Leavitt R, Snyder S, McAuliffe V, Boucher C. Baseline human immunodeficiency virus type 1 phenotype, genotype, and RNA response after switching from long-term hard-capsule saquinavir to indinavir or soft-gel-capsule saquinavir in AIDS clinical trials group protocol 333. J Infect Dis. 2000 Sep;182(3):733-43. doi: 10.1086/315769. Epub 2000 Aug 14. PMID 10950766